CLINICAL TRIAL: NCT02928432
Title: Phase II Pilot Study of the Prednisone to Dexamethasone Switch in Metastatic Castration Resistant Prostate Cancer (CRPC) Patients With Asymptomatic Biochemical and/or Limited Radiological Progression on Abiraterone and Prednisone
Brief Title: SWITCH: Study of the Prednisone to Dexamethasone Change in mCRPC Patients Treated With Abiraterone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Instituto de Investigacion Biomedica de Malaga (Other); Fundación de investigación HM (Other); Institute of Cancer Research, United Kingdom (Other); University of Salamanca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNIO-CP-05-2015
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Castration-Resistant Prostate Cancer; Abiraterone acetate; Steroids Switch
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: One-arm prospective
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Steroids switch (Experimental): CRPC patients with biochemical and/or limited radiological progression after at least 12 weeks of AA + prednisone.
  Interventions: Drug: Steroids switch

INTERVENTIONS:
Drug: Steroids switch — Change of prednisone 5mg/12h to dexamethasone 0.5mg/24h

SUMMARY:
Abiraterone acetate (AA) has shown a favourable impact in overall survival, administered with prednisone to decrease the adverse event related to CYP171A suppression.

Our hypothesis is that the change of prednisone to dexamethasone in CRPC patients that progress biochemically to AA + prednisone can improve the number and the length of the responses, and also improve tolerance to treatment, decreasing the adverse events associated to a moderate dosage of steroids used chronically.

DETAILED DESCRIPTION:
This phase II multicentric-study analyse the role of the steroid switch in patients receiving AA. Previous retrospective data (Lorente et al, BJC 2014) has shown that the change of prednisone by dexamethasone in CRPC patients treated with AA post-docetaxel leaded to durable biochemical responses in 40% of cases. Recently, superiority of dexamethasone over prednisone in PSA response has been reported by a phase II trial that included 82 chemotherapy-naive metastatic CRPC patients.

In our study patients with biochemical and/or limited radiological progression to AA + prednisone are prospectively enrolled. The principal objective was to evaluate the percentage of PSA responses in clinically stable metastatic CRPC patients after at least 12 weeks of AA + prednisone. Secondary aims will include time to biochemical progression, time to first radiological progression, overall survival and the evaluation of the safety profile.

Biochemical response was monitored with PSA determinations every 4 weeks, and defined as a ≥ 30% decline in PSA from baseline, confirmed with a second reading. PSA progression was evaluated according to PCWG2 criteria. Radiological response was re-evaluated every 12-16 weeks using bone and CT-scan according to RECIST v1.1 and PCWG2 criteria.

Translational studies: archival tissue will be obtained from all patients, to perform PTEN and TMPRSS-ERG rearrangements evaluation. Plasma will be collected after AA + prednisone progression to study the androgen receptor status in plasma.

ELIGIBILITY:
INCLUSION CRITERIA

1. Provision of signed informed consent
2. Patients must be 18 years old or older
3. Patients must have an acceptable performance status at study entry ECOG <2, without prior deterioration due to disease clinical progression on abiraterone plus prednisone
4. Patients must have prior histological confirmation of prostate cancer diagnosis prior to study entry
5. Maintained castration status to LHRH analogs/antagonist or surgical castration with Testosterone blood levels <0.5ng/mL should have been documented before the initiation of prior abiraterone plus prednisone treatment and confirmed again at study entry. Patients on LHRHa must be able to continue on them through the duration of the study.
6. Biochemical progression to abiraterone plus prednisone is required before study entry. This progression will be documented by a rising PSA value with an increase ≥25% and >2ng/dL over nadir, and must be confirmed by a second determination at least 2 weeks later should be documented before study entry.
7. Candidates must be able to swallow pills and to continue with abiraterone acetate dose of 1000mg/24h and must not have any contraindication for dexamethasone use at 0.5 mg/24h.
8. Patients must be asymptomatic or do not have any symptomatic deterioration attributable to prostate cancer progression at study entry
9. Absence of significant radiological progression to abiraterone plus prednisone at study entry. Only those cases with limited progression will be eligible if: a) they have not developed any new visceral, nodal or other soft tissue metastases; b) their measurable target lesions on abiraterone plus prednisone according to RECIST 1.1 should have not increased more than 40% from baseline or from their best response on treatment measurements; and c) they must have < 3 new bone metastasis on bone-scan from baseline according to PCWG2
10. Acceptable hematological, hepatic and renal functions, without contraindications for the administration of abiraterone: a) WBC count >2000/mm^3; b) Haemoglobin level >10 g/dL; c) Platelets >75000/mm^3; AST/ALT <2.5 times the upper normal limit; Total bilirubin <1.5 times the upper normal limit; Creatinine value <1.5 times the upper normal limit or creatinine clearance >50 ml/min

EXCLUSION CRITERIA

1. Any medical contraindication to continue on abiraterone acetate or to receive continuous daily low-dose of dexamethasone (0.5 mg/24h)
2. Any event which is considered clinical progression to abiraterone acetate by the attending physicians in the investigators team.
3. Any skeletal symptomatic event related to prostate cancer progression on abiraterone-acetate, except the administration of external beam radiotherapy due to bone-metastasis related-pain in a single area and which have resulted in a adequate symptom control for at least 4-weeks before study entry.
4. Radiological progression: a) New nodal, visceral or other soft tissue metastasis during the treatment with Abiraterone acetate and prednisone; b) increase of any target lesion >40% according to RECIST v1.1 criteria; c) any known visceral, nodal or soft tissue metastasis localisation causing symptomatic progression, and d) ≥ 3 new bone metastasis on bone-scan during treatment with abiraterone plus prednisone.
5. Previous cancer diagnosis, except those patients who had a localized malignant tumour and who are five years cancer-free, as well as subjects with a history of skin cancers (of non-melanoma type) or excised in situ carcinomas.
6. Any prior medical history, be they psychiatric or of any other character, which, according to the judgement of the investigator, might interfere with the subject's granting of informed consent or the safe execution of the procedures required in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the percentage of PSA response in metastatic CRPC treated with AA + dexamethasone with biochemical and/or limited radiological progression. | 12 months
  Biochemical response will be defined as a ≥ 30% decline in PSA from starting AA + dexamethasone, confirmed with a second PSA reading at least 2 weeks apart.

SECONDARY OUTCOMES:
To study time to biochemical (PSA) progression (>25% increase over PSA nadir value)in metastatic CRPC treated with AA + dexamethasone with biochemical and/or limited radiological progression. | 12 months
  Time to biochemical progression is defined as the time from AA + dexamethasone starting data, to PSA progression according to PCWG2 criteria
To analyze the time to radiological progression in metastatic CRPC treated with AA + dexamethasone with biochemical and/or limited radiological progression. | 24 months
  Time to radiological progression is defined as the time from AA+ dexamethasone starting date to the first occurrence of either progression by bone scan or progression by CT-scan (based on RECIST v1.1 and PCWG2 criteria), or death resulting from any cause.
To evaluate the overall survival in metastatic CRPC treated with AA + dexamethasone with biochemical and/or limited radiological progression. | 24 months
  Overall survival is defined as the time from AA + dexamethasone starting date to the death or last follow up visit.
To report the safety profile in in metastatic CRPC treated with AA + dexamethasone with biochemical and/or limited radiological progression. | 24 months
  Toxicity events will be collected prospectively in each visit according to CTCAE v4.0 criteria.
To describe the activity of subsequent treatment-line after AA + dexamethasone in the study population. | 24 months
  Subsequent therapies and their corresponding biochemical/radiological responses will be also recorded.
To explore potential androgen receptor pathway related circulating- and tissue-biomarkers in in metastatic CRPC treated with AA + dexamethasone with biochemical and/or limited radiological progression. | 24 months
  Archival tissue for immunohistochemistry and FISH, and peripheral blood to extract plasma and perform AR amplification studies by ddPCR analysis and determination of AR Alternative splicing transcripts from exosomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Spanish National Cancer Research Centre (CNIO), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No